CLINICAL TRIAL: NCT02195713
Title: Evaluation of a Novel Electronic Urine Output Monitor (eUOM)
Status: Completed | Type: Observational
Sponsor: Potrero Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: PM-JMSRF2014-BCF01
Record Dates: First submitted 2014-07-15; First posted 2014-07-21 (Estimated); Results first posted 2015-09-01 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-01

CONDITIONS: Oliguria; Polyuria
MeSH Terms: conditions — Oliguria; Polyuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Test- Accuryn Urine Output Monitor: Accuryn Anti-airlock Drainage System was attached to the Foley catheter and urine output / drainage line pressure was monitored.
  Interventions: Device: Accuryn
- Control- Critcore Urine Output Monitor: A commercially available urine output monitor (Criticore, Bard Medical) was attached to the Foley catheter and urine output / drainage line pressure was monitored.

INTERVENTIONS:
Device: Accuryn — Accuryn is a novel electronic urine output monitor
  Groups: Test- Accuryn Urine Output Monitor

SUMMARY:
Urine output and urine drain line pressure were monitored while urine was drained into either:

1. Accuryn Urine Output Monitor (Potrero Medical) OR
2. Criticore Monitor (Bard Medical)

DETAILED DESCRIPTION:
The purpose of this study is to determine the characteristics of urine output and drain line pressure as measured with the Accuryn urinary output monitoring system and urine output as recorded by a commercially available system (Criticore, Bard Medical) when used with a standard Foley catheter and standard urinary drainage tube.

ELIGIBILITY:
Inclusion Criteria:

* Patient must ≥ 18 years of age
* Patient has a Foley catheter and urine collection system is in place per standard clinical decision
* Estimated length of placement of the Foley is 48 hours minimum
* Burn injury ≥ 20% and ≤ 80% total body surface area (TBSA)
* Subject or subject's legally authorized representative is able to give informed consent before entering the study

Exclusion Criteria:

* Currently pregnant or breastfeeding
* Clinical signs or symptoms of a urinary tract infection (UTI)
* Clinical signs or symptoms of a vaginal infection
* Currently has bladder or urethral trauma
* Use of investigational drug/device therapy within the past 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patient that needs a Foley catheter
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-07; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Kramer, Principal Investigator — UTMB; Bruce Friedman, Principal Investigator — Joseph M. Stills Burn Center
Locations (2):
- United States (2):
  - Joseph M. Still Burn Center at Doctors Hospital, Augusta, Georgia
  - The University of Texas Medical Branch (UTMBP), Galveston, Texas

REFERENCES:
- See also: Related Info — http://potreromed.com

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Test- Accuryn Urine Output Monitor | Control- Critcore Urine Output Monitor
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test- Accuryn Urine Output Monitor | Control- Critcore Urine Output Monitor | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (22) | 52 (17.9) | 49 (20.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 7 | 8 | 15
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Urine Output of SOC Device Versus Accuryn
Description: Urine output as recorded by the SOC when connected to a standard Foley catheter and standard urinary drainage tube will be compared to urine output recorded by Accuryn and the SOC when connected to a standard Foley catheter and the Accuryn Drainage Tube.
Time Frame: 2 - 5 days
Measure: Number (95% Confidence Interval); unit: Patients with airlocks
Arm/Group | Test- Accuryn Urine Output Monitor | Control- Critcore Urine Output Monitor
Number analyzed (Participants) | 10 | 10
Patients with airlocks | 0 [0 to 0] | 5 [5 to 5]

ADVERSE EVENTS:
Arm/Group | Test- Accuryn Urine Output Monitor | Control- Critcore Urine Output Monitor
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No